CLINICAL TRIAL: NCT00531778
Title: NYU Ovarian Cancer Early Detection Program Blood and Genetics
Status: Terminated | Type: Observational
Why Stopped: insufficient funding and resource
Sponsor: NYU Langone Health (Other)
Responsible Party: Bhavana Pothuri, M.D., NYU Cancer Institute
Other Study IDs: NYU 04-30 H11938
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Ovarian Cancer
Keywords: Women with increased risk for developing ovarian cancer; early detection; biomarker for ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, urine, ovarian tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NYU OCEDP Population

SUMMARY:
Improving current strategies for detection of early stage disease can impact favorably on long-term survival of women with ovarian cancer. To reduce the morbidity and mortality of ovarian cancer, screening for this disease must detect early stage disease rather than advanced stage disease. Thus the challenge for the future is to identify and develop highly sensitive and specific tumor markers that can be applied to population-based screening for the early detection of ovarian cancer.

DETAILED DESCRIPTION:
The aim of NYU Ovarian Cancer Early Detection Program is to establish an effective, early detection program employing state-of-the-art science and technology in collaboration with other nationally recognized clinicians and scientists.

This proposed research study will foster collaboration between clinicians and scientists that will facilitate the rapid identification of a set of molecular, biochemical, functional, and genetic markers which can be employed to effectively detect and manage ovarian cancer and other gynecological malignancies.

ELIGIBILITY:
Inclusion Criteria:

Women enrolled in the NYU Ovarian Cancer Early Detection Program have at least one of the following risk factors:

* A personal history of breast cancer
* One or more first degree relatives (mother, sister, daughter) with ovarian cancer
* Multiple family members with either breast and/or ovarian cancer
* A personal history of a positive BRCA1 or BRCA2 genetic test result
* A close relative with a positive BRCA1 or BRCA2 genetic test result
* A personal history of colon or endometrial cancer with at least two relatives with a Lynch/HNPCC-associated cancer (colorectal, endometrial, small bowel, ureter, or renal pelvis cancer)
* Synchronous or metachronous endometrial and colorectal cancer
* A personal history of a mismatch repair gene mutation (MLH1, MSH2, MSH6 or PMS2)
* A close relative with a mismatch repair gene mutation (MLH1, MSH2, MSH6 or PMS2)
* A personal history of colorectal or endometrial cancer with a mismatch repair defect (ie. Microsatellite instability (MSI) or immunohistochemical loss of expression of MLH1, MSH2, MSH6, or PMS2)
* The use of fertility drugs for more than one year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women noted to be at increased risk for developing ovarian cancer
Sampling Method: Probability Sample
Enrollment: 890 (Actual)
Dates: Start 2004-06; Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
identification and development of highly sensitive and specific tumor markers for ovarian cancer | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Pothuri, M.D., Principal Investigator — NYU Langone Health
Locations (1):
- NYUCancer Institute Clinical Cancer Center, New York, New York, United States